CLINICAL TRIAL: NCT06699082
Title: Effects of Kinesiotaping With Kaltenborn Mobilization on the Rate of Recovery in Freezing Stage of Adhesive Capsulitis
Brief Title: Kinesiotaping With Kaltenborn Mobilization Effects on Adhesive Capsulitis Recovery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Neelo Gul
Record Dates: First submitted 2024-09-12; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: Kinesiotaping; Kaltenborn mobilization; Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: Experimental Group: kinesiotaping along with Kaltenborn mobilization AP and PA glides Experimental group was treated with kinesiotaping along with Kaltenborn mobilization AP and PA glides. The treatment protocol was administered in 10 reps' and 3 sets.
  AP Glide and PA Glide were applied. Kinesiotaping: First the deltoid area was dried and cleansed, excessive hair were trimmed, the KT was cut into Y-shape and I- shape was applied. The conventional therapy included; hot pacK, TENS for 5 mins and AROMS exercises 10 reps 2 sets. Home plan exercises included pendulum exercise, towel stretch exercise, finger ladder exercises and cross body adduction exercise.
Who Masked: Participant
Masking Description: Control Group: Kaltenborn mobilization AP and PA glides 10 reps' x 3 sets along with conventional therapy (hot pack for 10 mins, tens for 5 mins, AROMS exercises 10 reps 2 sets). Control was treated with Kaltenborn mobilization AP and PA glides 10 reps' x 3 sets along with conventional therapy that include; hot pack for 10 mins, tens for 5 mins, AROMS exercises 10 reps 2 sets. Home plane exercises included pendulum exercise, towel stretch exercise, and finger ladder exercise, cross body adduction exercise.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: 1 (Experimental): Experimental group was treated with kinesiotaping along with Kaltenborn mobilization AP and PA glides. The treatment protocol was administered in 10 reps' and 3 sets, and AP and PA glide were given.
  Kinesiotaping: First the deltoid area was dried and cleansed, excessive hair were trimmed, the KT was cut into Y-shape and I- shape, after that whole length of the thumb was used to stretch the tape for about 15% to 25% and then from 25% to 50%. The tape was rubbed vigorously for few seconds, heat activates glue. The whole procedure takes about 15 to 20 minutes.
  Interventions: Other: KinesioTaping and Keltonborn Mobilization
- Control Group: 2 (Active Comparator): Control was treated with Kaltenborn mobilization AP and PA glides along with conservative treatment and Home plane exercises.
  Interventions: Other: KinesioTaping and Keltonborn Mobilization

INTERVENTIONS:
Other: KinesioTaping and Keltonborn Mobilization — Experimental group was treated with kinesiotape and kaltenborn mobilization while the non experimental group was treated with conventional therapy along with kaltenborn mobilization.
  Other Names: Conventional Therapy with Keltonborn Mobilization

SUMMARY:
The purpose of the study is to determine the Effects of Kinesiotaping with Kaltenborn Mobilization on Rate of Recovery in Freezing Stage of Adhesive Capsulitis. A randomized control trial was conducted at Habib physiotherapy complex Peshawar and Pak physio rehabilitation Peshawar. The sample size was 34 calculated through open-epi tool. The participants were divided into two groups each having 17 participants. The study duration was six months. Consecutive sampling technique was used for the selection of subjects for the study that fulfills the eligibility criteria was included in the study. Block randomization was used to allocate subjects into interventional and control arms of the trial. The first two patients who fulfill the criteria were allocated to interventional arm and the next two patients were allocated in control arm till completion of the sample size for both the arms. Tools used in this study are Goniometer, SPADI, NPRS. Data was collected before and immediately after the application of interventions. Data analyzed through SPSS version 20

DETAILED DESCRIPTION:
Human kinematics is always in spotlight and considered as a unique feature in which shoulder joint kinematics have grabbed the attention of researchers. The complexity of the shoulder joint is evident from the literature. It is having high functional demands and wide range of motion than any other joint in the human body. It is balanced by stability and mobility provided by number of ligaments, capsule, labrum and active muscles. However sometimes this balance is disturbed that results in different musculoskeletal complaints and pathologies in which one of them is adhesive capsulitis (1).The exact cause of adhesive capsulitis remains controversial.

However calcific tendinitis, glenohumeral arthritis, acromioclavicular arthritis, dupuytrens, contractures, breast cancer, cardiac issues, autonomic neuropathy, stroke, cervical disc disorders, humeral fractures, hypoadrenalism, Parkinson's disease are some of the known causes (7). It can also occur as a sequalae of osteoarthritis, rheumatoid arthritis or joint dislocation and fracture (8). The evaluation of adhesive capsulitis starts from a thorough history and proceeding towards physical examination, clinical tests and radiographic techniques. The patient usually recalls a mild trauma or accident that has caused damage to the shoulder joint, as well as limited range of motion especially external rotation, sleep disturbance and pain on insertion of deltoid and unable to perform overhead activities (9). Physical examination exposes loss of natural swing of arm. Scapular dyskinesis is also noted in some cases. shoulder joint may be painful to touch and muscle atrophy can be present. Loss of ROM is seen (9). Fasting blood sugar is performed in patients having diabetes mellitus. Since inflammation is its feature so erythrocyte sedimentation rate is suggested. Some special tests are also positive in this condition that are Neer impingement sign and Hawkin's-Kneddy. These tests are positive due to capsular stretch and internal impingement that occurs in this condition simultaneously but due to adhesive capsulitis (10). Adhesive capsulitis can be diagnosed using imaging studies like radiographs, magnetic resonance imaging, arthrography, ultrasound, and nuclear medicine. Magnetic resonance imaging is considered the gold standard due to its soft tissue visualization and scanning capabilities. However, some studies suggest that it may not accurately diagnose the condition due to the similar thickness of the Page 3 of 11 (Draft) coracohumeral ligament (10 11). Rahee Mulmulay and Himanshu Pathak et al describes kinesiotaping along with Kaltenborn mobilization and Kaltenborn mobilization alone on pain, range of motion and functional disability in patients with adhesive capsulitis is effective treatment to significant improvement in terms of pain, range of motion and functional disability (12). Literature review: A systematic and evidence based search of relevant literature was performed by utilizing PubMed and Google Scholar as search engines and the key words used were Kinesiotaping, mobilization, Kaltenborn mobilization, adhesive capsulitis, frozen shoulder conventional physical therapy, freezing stage. The purpose of the literature review is to find out the pre-existing literature regarding the Kinesiotaping with Kaltenborn mobalization effects on adhesive capsulitis recovery. In 2017 a randomized controlled trial conducted by Rahee Mulmulay and Himanshu Pathak et al on effectiveness of kinesiotaping along with kaltenborn mobilization and kaltenborn mobilization alone on pain, range of motion and functional disability in patients with adhesive capsulitis stated that there is significance improvement in terms of pain, range of motion and functional disability (12). In 2019 a randomized controlled trial conducted by Sumit Raghav et in India on effectiveness of Mulligan versus Kaltenborn mobilization in the management of adhesive capsulitis. The results of the study showed significant improvement in terms of pain, range of motion and functional disability (13).

ELIGIBILITY:
Inclusion Criteria:

* Both genders male and female.
* Age 35-60 years.
* Acute shoulder pain (10 to 36 weeks).
* Patients with diabetes mellitus.
* Referred and diagnose patients

Exclusion Criteria:

* Any fracture related to the shoulder joint.
* Post operative case and osteoporotic.
* Shoulder with manipulation under anesthesia.
* Steroid injection therapy
* Diagnosed rheumatoid arthritis
* Neurological deficits / Hemiplegics

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-08-29 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Numerical pain rating scale | 3 times a week for 3 weeks
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a unidimensional measure of pain intensity in adults,[1][2][3] including those with chronic pain due to rheumatic diseases The 11-points of numeric pain rating scale ranges from '0' representing one with no pain, 1 to 3 with mild pain, 4 to 7 with moderate pain and 8 to 10 representing the pain extreme.
shoulder pain and disability index | 3 times a week for 3 weeks
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.
Goniometry | 3 times a week for 3 weeks
  A goniometer is a device that measures an angle or permits the rotation of an object to a definite position. In orthopedics, the former description applies more. The art and science of measuring the joint ranges in each joint plane are called goniometry.
  Goniometric measurements were obtained by aligning the goniometer arms with bony landmarks and aligning the fulcrum of the goniometer with the approximate location of the glenohumeral joint axis.

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsu JE, Anakwenze OA, Warrender WJ, Abboud JA. Current review of adhesive capsulitis. J Shoulder Elbow Surg. 2011 Apr;20(3):502-14. doi: 10.1016/j.jse.2010.08.023. Epub 2010 Dec 16. No abstract available. PMID 21167743
- [Background] Cohen C, Ejnisman B. Epidemiology of frozen shoulder. Shoulder stiffness: Springer; 2015. p. 21-30.
- [Background] Kingston K, Curry EJ, Galvin JW, Li X. Shoulder adhesive capsulitis: epidemiology and predictors of surgery. J Shoulder Elbow Surg. 2018 Aug;27(8):1437-1443. doi: 10.1016/j.jse.2018.04.004. Epub 2018 May 25. PMID 29807717
- [Background] Gaspar PD, Willis FB. Adhesive capsulitis and dynamic splinting: a controlled, cohort study. BMC Musculoskelet Disord. 2009 Sep 7;10:111. doi: 10.1186/1471-2474-10-111. PMID 19735563
- [Background] White D, Choi H, Peloquin C, Zhu Y, Zhang Y. Secular trend of adhesive capsulitis. Arthritis Care Res (Hoboken). 2011 Nov;63(11):1571-5. doi: 10.1002/acr.20590. PMID 22034118
- [Background] Malavolta EA, Gracitelli MEC, Ribeiro Pinto GM, Freire da Silveira AZ, Assuncao JH, Ferreira Neto AA. Asian ethnicity: a risk factor for adhesive capsulitis? Rev Bras Ortop. 2018 Feb 23;53(5):602-606. doi: 10.1016/j.rboe.2018.02.004. eCollection 2018 Sep-Oct. PMID 30258826
- [Background] Wang K, Ho V, Hunter-Smith DJ, Beh PS, Smith KM, Weber AB. Risk factors in idiopathic adhesive capsulitis: a case control study. J Shoulder Elbow Surg. 2013 Jul;22(7):e24-9. doi: 10.1016/j.jse.2012.10.049. Epub 2013 Jan 24. PMID 23352186
- [Background] Robinson CM, Seah KT, Chee YH, Hindle P, Murray IR. Frozen shoulder. J Bone Joint Surg Br. 2012 Jan;94(1):1-9. doi: 10.1302/0301-620X.94B1.27093. PMID 22219239
- [Background] Struyf F, Meeus M. Current evidence on physical therapy in patients with adhesive capsulitis: what are we missing? Clin Rheumatol. 2014 May;33(5):593-600. doi: 10.1007/s10067-013-2464-3. Epub 2013 Dec 28. PMID 24374758
- [Background] Harris G, Bou-Haidar P, Harris C. Adhesive capsulitis: review of imaging and treatment. J Med Imaging Radiat Oncol. 2013 Dec;57(6):633-43. doi: 10.1111/1754-9485.12111. Epub 2013 Sep 10. PMID 24283550
- [Background] Song KD, Kwon JW, Yoon YC, Choi SH. Indirect MR arthrographic findings of adhesive capsulitis. AJR Am J Roentgenol. 2011 Dec;197(6):W1105-9. doi: 10.2214/AJR.10.6099. PMID 22109326
- [Background] Pathak RMaH. Effect Of Kinesiotaping Along With Kalternborn Mobilization In Patients With Sub Acute Adhesive Capsulitis. International Journal of Current Advanced Research. 2017;Vol 6(Issue 12):8489-98.
- [Background] Ragav S, Singh A. Comparison of Effectiveness of Mulligan ‗MWM'Technique versus Kaltenborn Mobilization Technique on Pain and End Range of Motion in Patients with Adhesive Capsulitis of Shoulder Joint: A Randomized Controlled Trial. Journal of Exercise Science & Physiotherapy Vol. 2019;15(1).